CLINICAL TRIAL: NCT03536676
Title: Benefits of a Higher Protein, 'Egg-cellent' Breakfast in the Classroom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17120035
Record Dates: First submitted 2018-05-02; First posted 2018-05-25 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Breakfast; Obesity; Mood; Eating Behavior
Keywords: Breakfast; Obesity; Mood; Eating Behavior; Cognitive Function
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional School Breakfast Program (Active Comparator): The breakfasts for the 3-week program will adhere to the United States Department of Agriculture nutrition requirements for Grades 6-8.
  Interventions: Other: Breakfast in the Classroom
- 'Egg-Cellent' Breakfast in the Classroom (Experimental): The breakfasts for the 3-week program will adhere to the United States Department of Agriculture nutrition requirements for Grades 6-8 but will include an additional 2 large eggs/breakfast.
  Interventions: Other: 'Egg-cellent' Breakfast in the Classroom

INTERVENTIONS:
Other: 'Egg-cellent' Breakfast in the Classroom — Includes the additional 2 eggs per day
  Arms: 'Egg-Cellent' Breakfast in the Classroom
Other: Breakfast in the Classroom — Receives the standard meal for Breakfast in the Classroom
  Arms: Traditional School Breakfast Program

SUMMARY:
This study will test whether whether the implementation of and Egg-cellent 'Breakfast in the Classroom' improves school breakfast participation and breakfast consumption in middle school adolescents; whether the implementation of 'Breakfast in the Classroom' improves appetite control, mood, cognitive performance, and unhealthy snacking behavior in middle school adolescents when compared to a traditional school breakfast program.

DETAILED DESCRIPTION:
The investigators propose an 4-week cross-over design breakfast study in children enrolled in 6-8th grade within the Center School District in the Kansas City, Missouri. This school will begin their 'Breakfast in the Classroom' program on March 26, 2018. Prior to the start of 'Breakfast in the Classroom', baseline data will be collected on the students who wish to participate in the study. Baseline data includes anthropometric assessments; demographics; current eating habits; cognitive performance; appetite; and mood. Following baseline, the students will be provided a breakfast that meets all the requirements for a reimbursable school breakfast with the addition of two eggs for 3-weeks: At 4 weeks (3 weeks after initiation of the program), the study participants will complete a similar outcomes to those completed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* All students from the Center Middle School in Kansas City, MO who choose to participate and whose parent/legal guardian (excluding Wards of the State) signs the consent will be included.

Exclusion Criteria:

* Wards of the State will be excluded from this study.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
School Breakfast Program Participation | 3-weeks prior to program initiation and 3-weeks of program
  Participation at during the traditional school breakfast program and throughout the Breakfast in the Classroom program will be determined by the electronic school meal tracking system that logs student participation each day for breakfast and lunch.

SECONDARY OUTCOMES:
Habitual Breakfast Habits Questionnaire | Baseline and 3-weeks after beginning the intervention
  During one day, a questionnaire assessing previous breakfast habits will be given to participants. This questionnaire asks how many days per week they consume various breakfast foods.
Benefits of Breakfast Questionnaire | Baseline and 3-weeks after beginning the intervention
  During one day, a questionnaire asking the participants what happens when participants consume breakfast and skip breakfast will be administered. They will be given a list of choices (multiple selections are allowed) and the units for analysis will be binary (they chose it or did not choose it).
Snacking Questionnaires | Baseline and 3-weeks after beginning the intervention
  During one day, questionnaires assessing typical snacking behavior will be completed once. Participants will be asked to think about what they ate during the past week. They will be asked how many times they ate a variety of foods throughout this week. The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available).
Cognitive Performance Assessment | Baseline and 3-weeks after beginning the intervention
  During one day, cognitive performance assessments will occur once between 120 min and 180 min after breakfast using the online CNS Vital Signs neurocognitive assessment system during one day. The CNS Vital Signs system contains a battery of computerized tests to assess attention, memory, executive function, and cognitive flexibility. The assessment will occur outside of classroom learning activities.
Appetite Questionnaires | Baseline and 3-weeks after beginning the intervention
  Questionnaires, assessing hunger, fullness, prospective food consumption, and eating initiation, will be completed during the following times for 1 day immediately before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Mood State Questionnaires | Baseline and 3-weeks (Post-study)
  Questionnaires assessing tiredness, sleepiness, energy, irritability/agitation, etc.) will be completed during the following times for 1 day immediately before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Breakfast in the Classroom Participation Questionnaire | Baseline and 3-weeks after beginning the intervention
  Questionnaires assessing whether they ate breakfast or skipped breakfast and what types of foods they ate (if they ate breakfast) will be completed for 5 consecutive days during baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Leidy, PhD, Principal Investigator — Associate Professor
Locations (1):
- Center Middle School, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No